CLINICAL TRIAL: NCT03715361
Title: AF Stroke Substudy SL-ECG Versus 12lead ECG
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-078
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: ECG; Atrial Fibrillation; ECG Hand-held Diagnostic Tool
Keywords: ECG measurement; AF-Stroke; Germany; Electrocardiogram
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients (500 patients ≤ ) who undergo out- or inpatient treatment and who did a 12lead-ECG measurement, repeat the procedure using the hand-held diagnostic tool (SL-ECG).
  Interventions: Diagnostic Test: SL-ECG
- Control Group: Fifty volunteers who did a 12lead-ECG measurement, repeat the procedure using the hand-held diagnostic tool (SL-ECG).
  Interventions: Diagnostic Test: SL-ECG

INTERVENTIONS:
Diagnostic Test: SL-ECG — additional SL-ECG measurement

SUMMARY:
The purpose of the study is to compare parameters obtained per SL-ECG with the values from 12lead-ECG measurement. Patients who undergo out- or inpatient treatment and who receive a 12lead-ECG are asked to participate in this examination. Furthermore, 50 patients without heart disease should be included (control group).

DETAILED DESCRIPTION:
Atrial fibrillation is the most common cardiac arrhythmia in Germany. Clinical studies have shown that atrial fibrillation is associated with increased morbidity and mortality and reduced quality of life. Patients with atrial fibrillation have a three times higher risk of heart failure and a four to five times higher risk of ischemic stroke. In addition to these risks, atrial fibrillation is often asymptomatic and therefore more difficult to diagnose. It is estimated that about one third of all atrial fibrillation patients are asymptomatic.

For this reason, the study "Opportunistic Screening in Pharmacies for Atrial Fibrillation in Seniors" was conducted in Aachen. Within four weeks more than 7000 volunteers could be measured in participating pharmacies using a ECG hand-held diagnostic tool. Since the already measured subjects only have the SL-ECG measurement of the hand-held diagnostic tool, the aim of this substudy is to establish a reference group. In this reference group a 12lead-ECG is performed by routine ECG and a SL-ECG measurement by ECG hand-held diagnostic tool. The aim of the study is to compare the measured parameters and to optimize the algorithm to evaluate the remaining SL-ECGs of the main study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years old, for minors the signature of the legal guardian is required.
* Understanding of the essence, meaning and scope of the study.
* Patients (in-/outpatient) who receive a 12lead ECG through Medical Clinic 1.
* Volunteers who are willing to have a 12lead ECG and an SL-ECG performed and provide medical information.
* Signed informed consent

Exclusion Criteria:

* Insufficient language skills
* Limited cognitive abilities
* Limited physical abilities (i.e. tremor)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients and volunteers that meets the inclusion criteria and are not affected by the exclusion criteria are allowed to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Comparison of the SL-ECG (hand-held diagnostic tool) with the 12lead-ECG (gold standard) to identify and evaluate cardiac arrhythmias. | 12 Month
  The 12lead-ECG and the measurement of the hand-held diagnostic tool, performed by the proband/volunteer after the main examination, are crucial for the examination. The ECG hand-held diagnostic tool measures the heartbeat by analyzing the RR-intervals and gives a direct indication of irregularities through a red light after the measurement. Preliminary analyses showed a very good signal quality of the SL-ECG, therefore the times [s] and amplitudes [mV] of the P-wave, QRS-complex, T-wave, as well as the conduction and excitation shall be compared with each other and evaluated.

SECONDARY OUTCOMES:
Analysis of SL-ECGs and validation of prognostic factors based person-specific data and their medical history. | 12 Month
  The descriptive analysis is performed comprehensively for the entire cohort and separately for people with known and newly discovered atrial fibrillation. The SL-ECG, person-specific data (e.g. age, BMI) and medical history (e.g. cardiovascular diseases, drug intake) are used to validate known prognostic factors and to find new prognostic factors. Continuous variables are summarized by calculating mean, median, standard deviation, quantiles and interquartile distances. For categorial variables, frequencies and percentages are calculated and tabulated. Based on these values, the raw incidence as well as age- and gender-specific incidences of atrial fibrillation can be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, Principal Investigator — Head of the Clinic for Cardiology, Pneumology, Angiology and Internal Intensive Medicine
Locations (1):
- Uniklinium RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Chugh SS, Blackshear JL, Shen WK, Hammill SC, Gersh BJ. Epidemiology and natural history of atrial fibrillation: clinical implications. J Am Coll Cardiol. 2001 Feb;37(2):371-8. doi: 10.1016/s0735-1097(00)01107-4. PMID 11216949
- [Background] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Background] Schnabel RB, Wilde S, Wild PS, Munzel T, Blankenberg S. Atrial fibrillation: its prevalence and risk factor profile in the German general population. Dtsch Arztebl Int. 2012 Apr;109(16):293-9. doi: 10.3238/arztebl.2012.0293. Epub 2012 Apr 20. PMID 22577476
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- See also: www.ahajournals.org/doi/abs/10.1161/CIRCULATIONAHA.114.014343 — http://onlinelibrary.wiley.com/doi/pdf/10.1111/j.1538-7836.2005.01344.x